CLINICAL TRIAL: NCT02986854
Title: A Phase 3b, Controlled, Open-Label, Multi-Center Study to Evaluate Safety and Immunogenicity of a Single Dose of GlaxoSmithKline's Meningococcal ACWY Conjugate Vaccine (Menveo), Administered to Healthy Individuals 15 Through 55 Years of Age, Approximately 4-6 Years After Primary ACWY Vaccination
Brief Title: Study to Assess the Safety and Immunogenicity of a Single Dose of GlaxoSmithKline's (GSK) Meningococcal MenACWY-CRM Vaccine (Menveo), Administered to Subjects 15 Through 55 Years of Age, Approximately 4-6 Years After Primary ACWY Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205352; V59_77 (Other: Novartis); 2016-003186-25 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal disease; Booster vaccination; Meningitis; Antibody persistence
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Menveo-Menveo Group (Experimental): Approximately 300 subjects, who were vaccinated with a single dose of Menveo 4 to 6 years before, will receive one dose of MenACWY-CRM at Day 1.
  Interventions: Biological: Meningococcal (groups A, C, W and Y) oligosaccharide diphtheria CRM-197 conjugate Vaccine (Menveo)
- Menactra-Menveo Group (Experimental): Approximately 300 subjects, who were vaccinated with a single dose of Menactra 4 to 6 years before, will receive one dose of MenACWY-CRM at Day 1.
  Interventions: Biological: Meningococcal (groups A, C, W and Y) oligosaccharide diphtheria CRM-197 conjugate Vaccine (Menveo)
- Naive Group (Active Comparator): Aproximately 100 subjects, of similar age to subjects enrolled in other primed groups, who have not received any meningococcal vaccination, will receive one dose of MenACWY-CRM at Day 1.
  Interventions: Biological: Meningococcal (groups A, C, W and Y) oligosaccharide diphtheria CRM-197 conjugate Vaccine (Menveo)

INTERVENTIONS:
Biological: Meningococcal (groups A, C, W and Y) oligosaccharide diphtheria CRM-197 conjugate Vaccine (Menveo) — One intramuscular injection of MenACWY at Day 1.

SUMMARY:
The purpose/aim of this study is to assess the safety and antibody response to vaccination with a booster dose of Menveo given 4-6 years after primary MenACWY vaccination and to assess the safety and antibody response to a single dose of Menveo given to vaccine-naïve subjects

DETAILED DESCRIPTION:
This is a phase 3b, controlled, open-label, multi-center study to evaluate safety and immunogenicity of Menveo after a single vaccination in healthy individuals who were vaccinated with Menveo or Menactra 4 to 6 years before and in vaccine-naive individuals. Vaccine-naive subjects: subjects who have not received any meningococcal vaccine prior to participation to this clinical trial.

Subjects will be randomised into one of the two different blood draw schedules according to a 1:1 ratio.

* Blood draws at Day 1, Day 4 and Day 29
* Blood draws at Day 1, Day 6 and Day 29

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 15 through 55 years of age on the day of informed consent or assent.
2. Individuals who received Menveo 4 to 6 years prior to enrolment at an age of 11 years or older OR Individuals who received Menactra 4 to 6 years prior to enrolment at an age of 11 years or older OR Individuals who have not received any previous meningococcal vaccine.
3. Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry. If the subject is under age 18 at the time of enrolment, the parent(s)/legal guardian(s) of the subject should have voluntarily given written informed consent.
4. Individuals who can comply with study procedures including follow-up.
5. Males Or Females of non-childbearing potential Or

   * Females of childbearing potential who are using an effective birth control method which they intend to use for at least 30 days after the study vaccination.

Exclusion Criteria:

Each subject must not have:

1. History of any meningococcal vaccine administration other than the single vaccination given 4 to 6 years before OR History of any meningococcal vaccine administration.
2. Current or previous, confirmed or suspected disease caused by N. meningitidis.
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days prior to study vaccination.
4. Progressive, unstable or uncontrolled clinical conditions.
5. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
6. Clinical conditions representing a contraindication to intramuscular vaccination (IM) and blood draws.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to study vaccination.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to study vaccination.
8. Received immunoglobulins or any blood products within 180 days prior to informed consent.
9. Received systemic antibiotic treatment within 3 days prior to study vaccination or blood draw.
10. Received an investigational or non-registered medicinal product within 30 days prior to study vaccination.
11. Study personnel as an immediate family or household member.
12. Individuals who have received any other vaccines within 7 days or 14 days prior to vaccination in this study or who are planning to receive any vaccine within 28 days from the study vaccination.
13. Individuals who have experienced a moderate or severe acute infection and/or fever defined as a temperature ≥38°C (100.4°F) within 3 days prior to study vaccination.
14. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 704 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (30):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
- GSK Investigational Site, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20103

REFERENCES:
- [Background] Tipton M, Daly W, Senders S, Block SL, Lattanzi M, Mzolo T, Barbi S, Pellegrini M, Keshavan P. MenACWY-CRM conjugate vaccine booster dose given 4-6 years after priming: Results from a phase IIIb, multicenter, open label study in adolescents and adults. Vaccine. 2019 Sep 30;37(42):6171-6179. doi: 10.1016/j.vaccine.2019.08.065. Epub 2019 Sep 5. PMID 31495595
- See also: Full CSR posting on GSK — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=205352&attachmentIdentifier=4b9c0f0f-df12-453e-bed2-1e14b1b278a1&fileName=gsk-205352-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 center in Puerto Rico and 37 centers in Unites States.
Pre-assignment Details: 704 subjects were enrolled in this study. Out of the 704 enrolled, 701 received the study vaccine
Groups:
- Menveo-Menveo Group: Healthy subjects, 15 through 55 years of age were vaccinated with a single dose of Menveo (MenACWY-CRM) 4 to 6 years before and received one dose of MenACWY-CRM at Day 1.
- Menactra-Menveo Group: Healthy subjects,15 through 55 years of age were vaccinated with a single dose of Menactra (meningococcal diphtheria toxoid-conjugated MenACWY vaccine, MenACWY-D) 4 to 6 years before and received one dose of MenACWY-CRM at Day 1.
- Naive Group: Healthy subjects,15 through 55 years of age, who have not received any meningococcal vaccination, received one dose of MenACWY-CRM at Day 1.
Period: Overall Study
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Naive Group
Started | 301 | 300 | 100
Completed | 298 | 288 | 97
Not Completed | 3 | 12 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Menactra-Menveo Group: Healthy subjects, 15 through 55 years of age were vaccinated with a single dose of Menactra (meningococcal diphtheria toxoid-conjugated MenACWY vaccine, MenACWY-D) 4 to 6 years before and received one dose of MenACWY-CRM at Day 1.
- Total: Total of all reporting groups
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Naive Group | Total
Number analyzed (Participants) | 301 | 300 | 100 | 701
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.1 (3.66) | 17.9 (4.54) | 38.8 (10.47) | 20.5 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 156 | 68 | 368
  Male | 157 | 144 | 32 | 333
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 6 | 1 | 9
  Asian | 4 | 14 | 3 | 21
  Black or African American | 24 | 23 | 12 | 59
  Native Hawaiian or other Pacific Islander | 3 | 1 | 0 | 4
  Unspecified | 17 | 23 | 5 | 45
  White | 251 | 233 | 79 | 563

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Antibody (hSBA) Seroresponse Against Neisseria Meningitidis Serogroups A, C, W and Y.
Description: Seroresponse was defined as follows:for subjects with pre-vaccination hSBA titers< 4,postvaccination hSBA titers≥16;for subjects with pre-vaccination hSBA titers≥4,post vaccination hSBA titers of atleast 4 times the pre-vaccination titers.Criteria to demonstrate primary objectives:Immune response sufficiency was tested sequentially;first in the group of subjects who received primary vaccination with Menveo &,if met,also in group of subjects who received primary vaccination with Menactra.Immune response is considered sufficient if lower limit of the 1-sided 97.5% CI for percentage of subjects with hSBA seroresponse against serogroups A, C, W & Y is greater than 75%.Study is considered successful if immune response sufficiency is demonstrated atleast in group of subjects who received primary vaccination with Menveo.This outcome measure was assessed only on subjects from Menveo-Menveo & Menactra-Menveo groups.Data from pooled and Naive groups are presented as part of secondary objectives
Time Frame: At Day 29
Population: Analysis was performed on the per protocol set for immunogenicity, which included all randomized subjects who had no protocol deviations and were not excluded due to other reasons defined prior to unblinding/analysis who received the study vaccination & provided evaluable serum samples at Day 29 with results available for atleast one serogroup
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Pooled Group (Menveo-Menveo and Menactra-Menveo): Pooled subjects from both Menveo-Menveo and Menactra-Menveo Groups
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 571 | 93
Percentage of subjects
  hSBA-Men A, Pre < 4: number analyzed (Participants) | 246 | 234 | 480 | 85
  hSBA-Men A, Pre < 4 | 97.97 [95.32 to 99.34] | 97.01 [93.93 to 98.79] | 97.50 [95.67 to 98.70] | 64.71 [53.59 to 74.77]
  hSBA-Men A, Pre ≥ 4: number analyzed (Participants) | 43 | 48 | 91 | 8
  hSBA-Men A, Pre ≥ 4 | 88.37 [74.92 to 96.11] | 93.75 [82.8 to 98.69] | 91.21 [83.41 to 96.13] | 75.00 [34.91 to 96.81]
  hSBA-Men A, Total seroresponse: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men A, Total seroresponse | 96.54 [93.73 to 98.33] | 96.45 [93.58 to 98.29] | 96.50 [94.64 to 97.85] | 65.59 [55.02 to 75.14]
  hSBA-Men C, Pre < 4: number analyzed (Participants) | 85 | 103 | 188 | 43
  hSBA-Men C, Pre < 4 | 100 [95.75 to 100] | 100 [96.48 to 100] | 100 [98.06 to 100] | 55.81 [39.88 to 70.92]
  hSBA-Men C, Pre ≥ 4: number analyzed (Participants) | 203 | 177 | 380 | 50
  hSBA-Men C, Pre ≥ 4 | 93.6 [89.3 to 96.55] | 93.79 [89.15 to 96.86] | 93.68 [90.75 to 95.91] | 58.00 [43.21 to 71.81]
  hSBA-Men C, Total seroresponse: number analyzed (Participants) | 288 | 280 | 568 | 93
  hSBA-Men C, Total seroresponse | 95.49 [92.4 to 97.57] | 96.07 [93.08 to 98.02] | 95.77 [93.78 to 97.27] | 56.99 [46.31 to 67.22]
  hSBA-Men W, Pre < 4: number analyzed (Participants) | 52 | 58 | 110 | 33
  hSBA-Men W, Pre < 4 | 100 [93.15 to 100] | 100 [93.84 to 100] | 100 [96.70 to 100] | 54.55 [36.35 to 71.89]
  hSBA-Men W, Pre ≥ 4: number analyzed (Participants) | 237 | 223 | 460 | 59
  hSBA-Men W, Pre ≥ 4 | 94.94 [91.32 to 97.36] | 91.48 [87.01 to 94.79] | 93.26 [90.57 to 95.38] | 25.42 [14.98 to 38.44]
  hSBA-Men W, Total seroresponse: number analyzed (Participants) | 289 | 281 | 570 | 92
  hSBA-Men W, Total seroresponse | 95.85 [92.86 to 97.84] | 93.24 [89.64 to 95.88] | 94.56 [92.37 to 96.28] | 35.87 [26.13 to 46.54]
  hSBA-Men Y, Pre < 4: number analyzed (Participants) | 115 | 123 | 238 | 54
  hSBA-Men Y, Pre < 4 | 100 [96.84 to 100] | 97.56 [93.04 to 99.49] | 98.74 [96.36 to 99.74] | 55.56 [41.40 to 69.08]
  hSBA-Men Y, Pre ≥ 4: number analyzed (Participants) | 172 | 157 | 329 | 39
  hSBA-Men Y, Pre ≥ 4 | 94.77 [90.3 to 97.58] | 91.72 [86.26 to 95.52] | 93.31 [90.05 to 95.76] | 46.15 [30.09 to 62.82]
  hSBA-Men Y, Total seroresponse: number analyzed (Participants) | 287 | 280 | 567 | 93
  hSBA-Men Y, Total seroresponse | 96.86 [94.13 to 98.56] | 94.29 [90.89 to 96.7] | 95.59 [93.56 to 97.13] | 51.61 [41.01 to 62.11]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A-day 29-Total seroresponse (Menveo-Menveo vs. Naive); Test type: Other — Differences in percentages and associated 95% CIs between study groups were calculated using the Miettinen & Nurminen score method; Miettinen & Nurminen score method; Difference in percentages = 30.95, 95% CI 2-sided [21.76 to 41.25]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A-day 29-Total seroresponse (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 30.86, 95% CI 2-sided [21.66 to 41.17]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A-day 29-Total seroresponse (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 30.91, 95% CI 2-sided [21.89 to 41.12]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- DAY 29 : Total seroresponse (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 0.09, 95% CI 2-sided [-3.15 to 3.36]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C-day 29-Total seroresponse (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 38.50, 95% CI 2-sided [28.54 to 48.90]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C-day 29-Total seroresponse (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 39.08, 95% CI 2-sided [29.16 to 49.46]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C-day 29-Total seroresponse (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 38.79, 95% CI 2-sided [29.03 to 49.06]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C-DAY 29 : Total seroresponse (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = -0.59, 95% CI 2-sided [-4.12 to 2.92]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W-day 29-Total seroresponse (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 59.98, 95% CI 2-sided [49.49 to 69.32]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W-day 29-Total seroresponse (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 57.37, 95% CI 2-sided [46.71 to 66.88]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W-day 29-Total seroresponse (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 58.69, 95% CI 2-sided [48.32 to 67.94]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W-DAY 29 : Total seroresponse (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 2.61, 95% CI 2-sided [-1.17 to 6.62]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y-day 29-Total seroresponse (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 45.25, 95% CI 2-sided [35.11 to 55.47]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y-day 29-Total seroresponse (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 42.67, 95% CI 2-sided [32.34 to 53.04]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y-day 29-Total seroresponse (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 43.98, 95% CI 2-sided [33.92 to 54.14]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- DAY 29 : Total seroresponse (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Difference in percentages = 2.58, 95% CI 2-sided [-0.86 to 6.3]

2. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An AE can be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom , or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. An unsolicited adverse event is an adverse event that was not solicited using a subject diary and that was spontaneously communicated by a subject and/or parent(s)/legal guardian(s) who has signed the informed consent.
Time Frame: Within 30 minutes after vaccination
Population: Analysis was performed on the unsolicited safety set which included all subjects who provided informed consent and demographic and/or baseline screening assessments, regardless of the subject's randomization and treatment status in the study, received a subject ID and reported any unsolicited adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 301 | 300 | 601 | 100
Participants | 0 | 8 | 8 | 1

3. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic AEs
Description: Assessed solicited local symptoms were injection site pain, erythema, induration. Assessed solicited systemic symptoms were fatigue, headache, myalgia, arthralgia, loss of appetite, nausea, chills and fever [defined and measured by a body temperature ≥37.5 degrees Celsius (ºC)]. Threshold for Erythema and Induration: Grade 0 (<25 mm), Any (>= 25 mm)
Time Frame: From Day 1 (6 hours) through Day 7 after vaccination
Population: Analysis was performed on the solicited safety set which included all subjects who provided informed consent and demographic and/or baseline screening assessments, regardless of the subject's randomization and treatment status in the study, received a subject ID and reported any solicited adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 296 | 296 | 592 | 97
Participants
  Any Local symptom | 119 | 97 | 216 | 41
  Any Systemic symptom | 162 | 148 | 310 | 35
  Any Induration: number analyzed (Participants) | 286 | 286 | 572 | 92
  Any Induration | 15 | 9 | 24 | 8
  Any Erythema: number analyzed (Participants) | 286 | 287 | 573 | 92
  Any Erythema | 12 | 8 | 20 | 10
  Any Pain: number analyzed (Participants) | 292 | 296 | 588 | 97
  Any Pain | 114 | 96 | 210 | 40
  Any Nausea: number analyzed (Participants) | 294 | 294 | 588 | 97
  Any Nausea | 48 | 44 | 92 | 13
  Any Fatigue: number analyzed (Participants) | 295 | 296 | 591 | 97
  Any Fatigue | 113 | 110 | 223 | 19
  Any Myalgia: number analyzed (Participants) | 294 | 296 | 590 | 97
  Any Myalgia | 55 | 54 | 109 | 15
  Any Arthralgia: number analyzed (Participants) | 294 | 295 | 589 | 96
  Any Arthralgia | 44 | 38 | 82 | 13
  Any Headache: number analyzed (Participants) | 294 | 295 | 589 | 97
  Any Headache | 100 | 82 | 182 | 21
  Any loss of apetite: number analyzed (Participants) | 294 | 296 | 590 | 97
  Any loss of apetite | 37 | 46 | 83 | 6
  Any chills: number analyzed (Participants) | 294 | 295 | 589 | 97
  Any chills | 34 | 35 | 69 | 10
  Fever | 2 | 5 | 7 | 0

4. Secondary Outcome: Number of Subjects Reporting Other Indicators of Reactogenicity
Description: Assessed indicators of reactogenicity were use of analgesics/antipyretics for prophylaxis, use of analgesics/antipyretics for treatment, body temperature (described as 0.5 °C increments from ≥ 36.0ºC)
Time Frame: From Day 1 (6 hours) through Day 7 after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 296 | 296 | 592 | 97
Participants
  Analgesics/antipyretics for prophylaxis: number analyzed (Participants) | 294 | 295 | 589 | 96
  Analgesics/antipyretics for prophylaxis | 13 | 15 | 28 | 5
  Analgesics/antipyretics for treatment: number analyzed (Participants) | 293 | 295 | 588 | 96
  Analgesics/antipyretics for treatment | 18 | 24 | 42 | 10
  Body temperature (36.0 - 36.4 ºC) | 68 | 57 | 125 | 16
  Body temperature (36.5 - 36.9 ºC) | 135 | 141 | 276 | 45
  Body temperature (37.0 - 37.4 ºC) | 83 | 77 | 160 | 33
  Body temperature (37.5 - 37.9 ºC) | 6 | 9 | 15 | 3
  Body temperature (38.0 - 38.4 ºC) | 1 | 2 | 3 | 0
  Body temperature (38.5 - 38.9 ºC) | 1 | 3 | 4 | 0
  Body temperature (39.0 - 39.4 ºC) | 0 | 0 | 0 | 0
  Body temperature (39.5 - 39.9 ºC) | 0 | 0 | 0 | 0
  Body temperature (>=40ºC) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Subjects Reporting All Unsolicited AEs
Description: An AE can be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom , or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. An unsolicited adverse event was an adverse event that was not solicited using a subject diary and that was spontaneously communicated by a subject and/or parent(s)/legal guardian(s) who has signed the informed consent.
Time Frame: From Day 1 through Day 29 after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 301 | 300 | 601 | 100
Participants | 74 | 78 | 152 | 22

6. Secondary Outcome: Number of Subjects Reporting Medically-attended AEs (MAAEs), AEs Leading to Withdrawal and Serious AEs (SAEs)
Description: Medically attended AEs were defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider.
  SAE was defined as any untoward medical occurrence that at any dose resulted in: death, was life-threatening, required or prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly/or birth defect, an important and significant medical event that might not have been immediately life threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, might jeopardized the subject or might required intervention to prevent one of the other outcomes listed.
Time Frame: From Day 1 through Day 181 (entire study period)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 301 | 300 | 601 | 100
Participants
  Any MAAEs | 102 | 79 | 181 | 19
  Any AEs leading to withdrawal | 0 | 0 | 0 | 0
  Any SAEs | 3 | 2 | 5 | 3

7. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥8 Against N. Meningitidis Serogroup A
Description: For each study group and in the pooled group, percentages of subjects with hSBA titer ≥8 and associated two-sided 95%CIs were calculated.
Time Frame: At Day 1 (pre-vaccination), Day 4, Day 6 and Day 29
Population: Analysis was performed on per protocol set for immunogenicity, which included all randomized subjects who had no protocol deviations and were not excluded due to other reasons defined prior to unblinding/analysis, who received study vaccination and provided evaluable serum samples at each time point, with result available for at least 1 serogroup
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 572 | 93
Percentages of subjects
  hSBA-Men A ≥ 8, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men A ≥ 8, Day 1 | 12.46 [8.88 to 16.83] | 14.89 [10.95 to 19.59] | 13.66 [10.95 to 16.75] | 4.3 [1.18 to 10.65]
  hSBA-Men A ≥ 8, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men A ≥ 8, Day 4 | 11.11 [6.49 to 17.42] | 13.04 [7.92 to 19.83] | 12.06 [8.5 to 16.44] | 4.17 [0.51 to 14.25]
  hSBA-Men A ≥ 8, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men A ≥ 8, Day 6 | 53.42 [44.99 to 61.71] | 47.14 [38.66 to 55.75] | 50.35 [44.4 to 56.29] | 9.09 [2.53 to 21.67]
  hSBA-Men A ≥ 8, Day 29 | 98.62 [96.51 to 99.62] | 98.94 [96.92 to 99.78] | 98.78 [97.49 to 99.51] | 70.97 [60.64 to 79.92]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 8.16, 95% CI 2-sided [1.23 to 13.41]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between group differences in percentage = 10.59, 95% CI 2-sided [3.54 to 16.14]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 1- (Pooled Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between group differences in percentage = 9.36, 95% CI 2-sided [2.72 to 13.58]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between group differences in percentage = -2.44, 95% CI 2-sided [-8.17 to 3.24]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 6.94, 95% CI 2-sided [-3.57 to 14.15]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 8.88, 95% CI 2-sided [-1.77 to 16.52]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 7.89, 95% CI 2-sided [-2.34 to 13.48]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -1.93, 95% CI 2-sided [-9.84 to 5.82]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 44.33, 95% CI 2-sided [30.25 to 54.60]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 38.05, 95% CI 2-sided [23.93 to 48.58]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 41.26, 95% CI 2-sided [28.15 to 49.72]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 6.28, 95% CI 2-sided [-5.31 to 17.71]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 27.65, 95% CI 2-sided [19.25 to 37.65]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 27.97, 95% CI 2-sided [19.60 to 37.95]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 27.81, 95% CI 2-sided [19.50 to 37.76]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -0.32, 95% CI 2-sided [-2.56 to 1.86]

8. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥8 Against N. Meningitidis Serogroup C
Description: as for outcome 7
Time Frame: At day 1(pre-vaccination) , day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 281 | 571 | 93
Percentage of subjects
  hSBA-Men C ≥ 8, Day 1: number analyzed (Participants) | 288 | 281 | 569 | 93
  hSBA-Men C ≥ 8, Day 1 | 61.11 [55.22 to 66.77] | 53.74 [47.72 to 59.68] | 57.47 [53.29 to 61.57] | 33.33 [23.89 to 43.87]
  hSBA-Men C ≥ 8, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men C ≥ 8, Day 4 | 70.83 [62.68 to 78.1] | 60.14 [51.47 to 68.38] | 65.6 [59.74 to 71.13] | 43.75 [29.48 to 58.82]
  hSBA-Men C ≥ 8, Day 6: number analyzed (Participants) | 145 | 139 | 284 | 44
  hSBA-Men C ≥ 8, Day 6 | 87.59 [81.09 to 92.47] | 92.09 [86.28 to 95.98] | 89.79 [85.66 to 93.05] | 43.18 [28.35 to 58.97]
  hSBA-Men C ≥ 8, Day 29 | 100 [98.74 to 100] | 99.64 [98.03 to 99.99] | 99.82 [99.03 to 100] | 87.1 [78.55 to 93.15]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 27.78, 95% CI 2-sided [16.23 to 38.27]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 20.40, 95% CI 2-sided [8.78 to 31.03]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 24.14, 95% CI 2-sided [13.28 to 33.86]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 7.37, 95% CI 2-sided [-0.76 to 15.42]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 27.08, 95% CI 2-sided [11.04 to 42.14]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 16.39, 95% CI 2-sided [0.04 to 31.90]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 21.85, 95% CI 2-sided [6.73 to 36.11]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 10.69, 95% CI 2-sided [-0.42 to 21.60]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 44.40, 95% CI 2-sided [28.65 to 58.93]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 48.90, 95% CI 2-sided [33.45 to 63.13]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 46.61, 95% CI 2-sided [31.52 to 60.59]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -4.50, 95% CI 2-sided [-11.84 to 2.69]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 12.90, 95% CI 2-sided [7.53 to 21.22]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 12.55, 95% CI 2-sided [7.10 to 20.89]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 12.73, 95% CI 2-sided [7.34 to 21.05]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.36, 95% CI 2-sided [-0.96 to 1.99]

9. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥8 Against N. Meningitidis Serogroup W
Description: as for outcome 7
Time Frame: At day 1(pre-vaccination), day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 571 | 93
Percentage of subjects
  hSBA-Men W ≥ 8, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men W ≥ 8, Day 1 | 75.43 [70.05 to 80.29] | 76.95 [71.59 to 81.74] | 76.18 [72.47 to 79.62] | 61.29 [50.62 to 71.22]
  hSBA-Men W ≥ 8, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men W ≥ 8, Day 4 | 81.94 [74.67 to 87.85] | 82.61 [75.24 to 88.53] | 82.27 [77.3 to 86.54] | 62.5 [47.35 to 76.05]
  hSBA-Men W ≥ 8, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men W ≥ 8, Day 6 | 93.84 [88.62 to 97.14] | 97.86 [93.87 to 99.56] | 95.8 [92.79 to 97.81] | 63.64 [47.77 to 77.59]
  hSBA-Men W ≥ 8, Day 29: number analyzed (Participants) | 290 | 281 | 571 | 92
  hSBA-Men W ≥ 8, Day 29 | 100 [98.74 to 100] | 100 [98.7 to 100] | 100 [99.36 to 100] | 84.78 [75.79 to 91.42]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 14.14, 95% CI 2-sided [3.46 to 25.39]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 15.66, 95% CI 2-sided [5.00 to 26.89]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 14.89, 95% CI 2-sided [4.91 to 25.62]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -1.52, 95% CI 2-sided [-8.51 to 5.50]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.44, 95% CI 2-sided [5.25 to 34.83]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 20.11, 95% CI 2-sided [5.88 to 35.50]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.77, 95% CI 2-sided [6.53 to 34.58]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -0.66, 95% CI 2-sided [-9.67 to 8.40]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 30.20, 95% CI 2-sided [16.78 to 45.45]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 34.22, 95% CI 2-sided [21.29 to 49.20]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 32.17, 95% CI 2-sided [19.30 to 47.13]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -4.02, 95% CI 2-sided [-9.45 to 0.74]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 15.22, 95% CI 2-sided [9.28 to 23.95]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 15.22, 95% CI 2-sided [9.28 to 23.95]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 15.22, 95% CI 2-sided [9.28 to 23.94]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0, 95% CI 2-sided [-1.31 to 1.35]

10. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥8 Against N. Meningitidis Serogroup Y
Description: as for outcome 7
Time Frame: At day 1(pre-vaccination), day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 281 | 571 | 93
Percentage of subjects
  hSBA-Men Y ≥ 8, Day 1: number analyzed (Participants) | 287 | 281 | 568 | 93
  hSBA-Men Y ≥ 8, Day 1 | 54.01 [48.05 to 59.88] | 46.98 [41.02 to 52.99] | 50.53 [46.33 to 54.72] | 32.26 [22.93 to 42.75]
  hSBA-Men Y ≥ 8, Day 4: number analyzed (Participants) | 143 | 138 | 281 | 48
  hSBA-Men Y ≥ 8, Day 4 | 55.24 [46.71 to 63.56] | 55.8 [47.1 to 64.24] | 55.52 [49.5 to 61.42] | 33.33 [20.4 to 48.41]
  hSBA-Men Y ≥ 8, Day 6: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men Y ≥ 8, Day 6 | 85.52 [78.72 to 90.81] | 87.86 [81.27 to 92.76] | 86.67 [82.16 to 90.39] | 45.45 [30.39 to 61.15]
  hSBA-Men Y ≥ 8, Day 29 | 100 [98.74 to 100] | 99.64 [98.03 to 99.99] | 99.82 [99.03 to 100] | 77.42 [67.58 to 85.45]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 21.75, 95% CI 2-sided [10.19 to 32.25]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 14.72, 95% CI 2-sided [3.15 to 25.29]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 18.27, 95% CI 2-sided [7.44 to 27.92]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 7.03, 95% CI 2-sided [-1.20 to 15.17]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 21.91, 95% CI 2-sided [5.57 to 36.37]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.46, 95% CI 2-sided [6.05 to 37.00]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.18, 95% CI 2-sided [6.89 to 35.38]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -0.55, 95% CI 2-sided [-12.11 to 11.03]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 40.06, 95% CI 2-sided [24.26 to 54.95]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 42.40, 95% CI 2-sided [26.71 to 57.17]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 41.21, 95% CI 2-sided [26.12 to 55.55]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -2.34, 95% CI 2-sided [-10.41 to 5.73]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.58, 95% CI 2-sided [15.26 to 32.08]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.22, 95% CI 2-sided [14.86 to 31.74]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.41, 95% CI 2-sided [15.08 to 31.90]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥8-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.36, 95% CI 2-sided [-0.96 to 1.99]

11. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥16 Against N. Meningitidis Serogroup A
Description: For each study group and in the pooled group, percentages of subjects with hSBA titer ≥16 and associated two-sided 95%CIs were calculated.
Time Frame: At day 1(pre-vaccination), day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 572 | 93
Percentage of subjects
  hSBA-Men A ≥ 16, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men A ≥ 16, Day 1 | 8.3 [5.39 to 12.1] | 9.57 [6.4 to 13.62] | 8.93 [6.72 to 11.58] | 1.08 [0.03 to 5.85]
  hSBA-Men A ≥ 16, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men A ≥ 16, Day 4 | 8.33 [4.38 to 14.1] | 8.7 [4.57 to 14.7] | 8.51 [5.53 to 12.4] | 2.08 [0.05 to 11.07]
  hSBA-Men A ≥ 16, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men A ≥ 16, Day 6 | 45.89 [37.62 to 54.33] | 41.43 [33.17 to 50.05] | 43.71 [37.87 to 49.67] | 4.55 [0.56 to 15.47]
  hSBA-Men A ≥ 16, Day 29 | 98.28 [96.02 to 99.44] | 97.52 [94.95 to 99] | 97.9 [96.36 to 98.91] | 66.67 [56.13 to 76.11]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 7.23, 95% CI 2-sided [2.08 to 11.23]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 8.50, 95% CI 2-sided [3.28 to 12.74]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 7.86, 95% CI 2-sided [2.87 to 10.78]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -1.27, 95% CI 2-sided [-6.10 to 3.49]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 6.25, 95% CI 2-sided [-3.04 to 12.44]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 6.61, 95% CI 2-sided [-2.71 to 13.01]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 6.43, 95% CI 2-sided [-2.66 to 10.90]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -0.36, 95% CI 2-sided [-7.27 to 6.43]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 41.34, 95% CI 2-sided [28.85 to 50.63]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 36.88, 95% CI 2-sided [24.39 to 46.34]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 39.16, 95% CI 2-sided [27.61 to 46.33]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 4.46, 95% CI 2-sided [-7.04 to 15.83]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 31.61, 95% CI 2-sided [22.68 to 41.79]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 30.85, 95% CI 2-sided [21.85 to 41.08]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 31.24, 95% CI 2-sided [22.39 to 41.38]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.76, 95% CI 2-sided [-1.81 to 3.52]

12. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥16 Against N. Meningitidis Serogroup C
Description: Analysis was performed on per protocol set for immunogenicity, which included all randomized subjects who had no protocol deviations and were not excluded due to other reasons defined prior to unblinding/analysis, who received study vaccination and provided evaluable serum samples at each time point, with result available for at least 1 serogroup
Time Frame: At day 1(pre-vaccination) , day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 281 | 571 | 93
Percentage of subjects
  hSBA-Men C ≥ 16, Day 1: number analyzed (Participants) | 288 | 281 | 569 | 93
  hSBA-Men C ≥ 16, Day 1 | 47.22 [41.34 to 53.16] | 38.08 [32.38 to 44.04] | 42.71 [38.6 to 46.89] | 17.2 [10.17 to 26.43]
  hSBA-Men C ≥ 16, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men C ≥ 16, Day 4 | 54.17 [45.67 to 62.49] | 44.93 [36.46 to 53.62] | 49.65 [43.66 to 55.64] | 29.17 [16.95 to 44.06]
  hSBA-Men C ≥ 16, Day 6: number analyzed (Participants) | 145 | 139 | 284 | 44
  hSBA-Men C ≥ 16, Day 6 | 82.07 [74.84 to 87.94] | 81.29 [73.81 to 87.4] | 81.69 [76.69 to 86.01] | 31.82 [18.61 to 47.58]
  hSBA-Men C ≥ 16, Day 29 | 99.66 [98.09 to 99.99] | 99.64 [98.03 to 99.99] | 99.65 [98.74 to 99.96] | 69.89 [59.5 to 78.97]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 30.02, 95% CI 2-sided [19.55 to 38.83]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 20.87, 95% CI 2-sided [10.48 to 29.69]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 25.50, 95% CI 2-sided [15.79 to 33.21]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 9.14, 95% CI 2-sided [1.01 to 17.16]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 25.00, 95% CI 2-sided [8.82 to 38.90]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 15.76, 95% CI 2-sided [-0.44 to 29.86]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 20.48, 95% CI 2-sided [5.32 to 33.08]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 9.24, 95% CI 2-sided [-2.45 to 20.68]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 50.25, 95% CI 2-sided [34.09 to 63.67]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 49.48, 95% CI 2-sided [33.21 to 63.01]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 49.87, 95% CI 2-sided [34.42 to 62.60]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.77, 95% CI 2-sided [-8.30 to 9.92]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 29.76, 95% CI 2-sided [21.34 to 39.75]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 29.75, 95% CI 2-sided [21.32 to 39.74]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 29.76, 95% CI 2-sided [21.35 to 39.73]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.01, 95% CI 2-sided [-1.60 to 1.67]

13. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥16 Against N. Meningitidis Serogroup W
Description: as for outcome 11
Time Frame: At day 1(pre-vaccination), day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 571 | 93
Percentage of subjects
  hSBA-Men W ≥ 16, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men W ≥ 16, Day 1 | 65.74 [59.96 to 71.2] | 66.31 [60.47 to 71.81] | 66.02 [61.98 to 69.91] | 48.39 [37.89 to 58.99]
  hSBA-Men W ≥ 16, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men W ≥ 16, Day 4 | 68.75 [60.5 to 76.21] | 76.81 [68.87 to 83.57] | 72.7 [67.1 to 77.81] | 54.17 [39.17 to 68.63]
  hSBA-Men W ≥ 16, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men W ≥ 16, Day 6 | 89.04 [82.81 to 93.6] | 92.14 [86.38 to 96.01] | 90.56 [86.56 to 93.69] | 50 [34.56 to 65.44]
  hSBA-Men W ≥ 16, Day 29: number analyzed (Participants) | 290 | 281 | 571 | 92
  hSBA-Men W ≥ 16, Day 29 | 100 [98.74 to 100] | 100 [98.7 to 100] | 100 [99.36 to 100] | 80.43 [70.85 to 87.97]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 17.36, 95% CI 2-sided [5.85 to 28.67]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 17.92, 95% CI 2-sided [6.39 to 29.25]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 17.64, 95% CI 2-sided [6.85 to 28.28]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -0.57, 95% CI 2-sided [-8.32 to 7.20]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 14.58, 95% CI 2-sided [-0.98 to 30.38]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 22.64, 95% CI 2-sided [7.30 to 38.16]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 18.53, 95% CI 2-sided [4.14 to 33.37]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -8.06, 95% CI 2-sided [-18.34 to 2.38]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 39.04, 95% CI 2-sided [23.76 to 54.07]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 42.14, 95% CI 2-sided [27.08 to 56.98]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 40.56, 95% CI 2-sided [25.91 to 55.15]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = -3.10, 95% CI 2-sided [-10.20 to 3.89]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.57, 95% CI 2-sided [12.74 to 28.83]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.57, 95% CI 2-sided [12.74 to 28.83]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.57, 95% CI 2-sided [12.75 to 28.83]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0, 95% CI 2-sided [-1.31 to 1.35]

14. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥16 Against N. Meningitidis Serogroup Y
Description: as for outcome 11
Time Frame: At day 1(pre-vaccination) , day 4, day 6 and day 29
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 281 | 571 | 93
Percentage of subjects
  hSBA-Men Y ≥ 16, Day 1: number analyzed (Participants) | 287 | 281 | 568 | 93
  hSBA-Men Y ≥ 16, Day 1 | 39.02 [33.35 to 44.93] | 34.88 [29.31 to 40.76] | 36.97 [32.99 to 41.09] | 17.2 [10.17 to 26.43]
  hSBA-Men Y ≥ 16, Day 4: number analyzed (Participants) | 143 | 138 | 281 | 48
  hSBA-Men Y ≥ 16, Day 4 | 39.16 [31.11 to 47.67] | 39.13 [30.94 to 47.8] | 39.15 [33.4 to 45.12] | 20.83 [10.47 to 34.99]
  hSBA-Men Y ≥ 16, Day 6: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men Y ≥ 16, Day 6 | 80.69 [73.31 to 86.77] | 80 [72.41 to 86.28] | 80.35 [75.26 to 84.8] | 31.82 [18.61 to 47.58]
  hSBA-Men Y ≥ 16, Day 29 | 100 [98.74 to 100] | 98.58 [96.4 to 99.61] | 99.3 [98.22 to 99.81] | 64.52 [53.91 to 74.17]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 21.82, 95% CI 2-sided [11.44 to 30.60]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 1- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 17.67, 95% CI 2-sided [7.34 to 26.43]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 1- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 19.77, 95% CI 2-sided [10.09 to 27.43]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 1- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 4.15, 95% CI 2-sided [-3.80 to 12.04]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 18.33, 95% CI 2-sided [2.92 to 30.99]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 4- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 18.30, 95% CI 2-sided [2.83 to 31.06]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 4- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 18.31, 95% CI 2-sided [3.83 to 29.39]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 4- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.03, 95% CI 2-sided [-11.35 to 11.39]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 48.87, 95% CI 2-sided [32.64 to 62.38]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 6- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 48.18, 95% CI 2-sided [31.87 to 61.79]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 6- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 48.53, 95% CI 2-sided [33.04 to 61.31]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 6- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 0.69, 95% CI 2-sided [-8.60 to 10.04]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 35.48, 95% CI 2-sided [26.50 to 45.62]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 29- (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 34.06, 95% CI 2-sided [24.94 to 44.28]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 29- (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 34.78, 95% CI 2-sided [25.78 to 44.93]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- hSBA titer ≥16-Vaccine comparison at Day 29- (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Between groups differences in percentage = 1.42, 95% CI 2-sided [0.10 to 3.60]

15. Secondary Outcome: Percentages of Subjects With hSBA Seroresponse Against N. Meningitidis Serogroups A, C, W and Y
Description: Seroresponse is defined for this study as follows: For subjects with pre-vaccination titers <4, postvaccination titers ≥ 16; for subjects with pre-vaccination titers ≥4, post vaccination titers at least 4 times the pre-vaccination titers.
Time Frame: At Day 4 and Day 6
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 289 | 282 | 571 | 93
Percentages of subjects
  hSBA-Men A, Pre < 4, Day 4: number analyzed (Participants) | 123 | 117 | 240 | 45
  hSBA-Men A, Pre < 4, Day 4 | 0.81 [0.02 to 4.45] | 2.56 [0.53 to 7.31] | 1.67 [0.46 to 4.21] | 0 [0 to 7.87]
  hSBA-Men A, Pre ≥ 4, Day 4: number analyzed (Participants) | 21 | 21 | 42 | 3
  hSBA-Men A, Pre ≥ 4, Day 4 | 4.76 [0.12 to 23.82] | 0 [0 to 16.11] | 2.38 [0.06 to 12.57] | 0 [0 to 70.76]
  hSBA-Men A, Total seroresponse, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men A, Total seroresponse, Day 4 | 1.39 [0.17 to 4.93] | 2.17 [0.45 to 6.22] | 1.77 [0.58 to 4.09] | 0 [0 to 7.4]
  hSBA-Men A, Pre < 4, Day 6: number analyzed (Participants) | 123 | 113 | 236 | 39
  hSBA-Men A, Pre < 4, Day 6 | 39.84 [31.12 to 49.05] | 33.63 [25.01 to 43.12] | 36.86 [30.7 to 43.37] | 2.56 [0.06 to 13.48]
  hSBA-Men A, Pre ≥ 4, Day 6: number analyzed (Participants) | 22 | 27 | 49 | 5
  hSBA-Men A, Pre ≥ 4, Day 6 | 36.36 [17.2 to 59.34] | 22.22 [8.62 to 42.26] | 28.57 [16.58 to 43.26] | 20 [0.51 to 71.64]
  hSBA-Men A, Total seroresponse, Day 6: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men A, Total seroresponse, Day 6 | 39.31 [31.31 to 47.76] | 31.43 [23.85 to 39.81] | 35.44 [29.89 to 41.3] | 4.55 [0.56 to 15.47]
  hSBA-Men C, Pre < 4, Day 4: number analyzed (Participants) | 36 | 51 | 87 | 20
  hSBA-Men C, Pre < 4, Day 4 | 0 [0 to 9.74] | 9.8 [3.26 to 21.41] | 5.75 [1.89 to 12.9] | 5 [0.13 to 24.87]
  hSBA-Men C, Pre ≥ 4, Day 4: number analyzed (Participants) | 107 | 86 | 193 | 28
  hSBA-Men C, Pre ≥ 4, Day 4 | 3.74 [1.03 to 9.3] | 8.14 [3.34 to 16.05] | 5.7 [2.88 to 9.97] | 7.14 [0.88 to 23.5]
  hSBA-Men C, Total seroresponse, Day 4: number analyzed (Participants) | 143 | 137 | 280 | 48
  hSBA-Men C, Total seroresponse, Day 4 | 2.8 [0.77 to 7.01] | 8.76 [4.61 to 14.8] | 5.71 [3.3 to 9.11] | 6.25 [1.31 to 17.2]
  hSBA-Men C, Pre < 4, Day 6: number analyzed (Participants) | 49 | 51 | 100 | 23
  hSBA-Men C, Pre < 4, Day 6 | 65.31 [50.36 to 78.33] | 64.71 [50.07 to 77.57] | 65 [54.82 to 74.27] | 13.04 [2.78 to 33.59]
  hSBA-Men C, Pre ≥ 4, Day 6: number analyzed (Participants) | 95 | 88 | 183 | 21
  hSBA-Men C, Pre ≥ 4, Day 6 | 44.21 [34.02 to 54.77] | 38.64 [28.44 to 49.62] | 41.53 [34.31 to 49.03] | 9.52 [1.17 to 30.38]
  hSBA-Men C, Total seroresponse, Day 6: number analyzed (Participants) | 144 | 139 | 283 | 44
  hSBA-Men C, Total seroresponse, Day 6 | 51.39 [42.92 to 59.8] | 48.2 [39.65 to 56.83] | 49.82 [43.85 to 55.8] | 11.36 [3.79 to 24.56]
  hSBA-Men W, Pre < 4, Day 4: number analyzed (Participants) | 21 | 30 | 51 | 17
  hSBA-Men W, Pre < 4, Day 4 | 9.52 [1.17 to 30.38] | 30 [14.73 to 49.4] | 21.57 [11.29 to 35.32] | 11.76 [1.46 to 36.44]
  hSBA-Men W, Pre ≥ 4, Day 4: number analyzed (Participants) | 123 | 108 | 231 | 31
  hSBA-Men W, Pre ≥ 4, Day 4 | 1.63 [0.2 to 5.75] | 4.63 [1.52 to 10.47] | 3.03 [1.23 to 6.14] | 3.23 [0.08 to 16.7]
  hSBA-Men W, Total seroresponse, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men W, Total seroresponse, Day 4 | 2.78 [0.76 to 6.96] | 10.14 [5.66 to 16.44] | 6.38 [3.83 to 9.9] | 6.25 [1.31 to 17.2]
  hSBA-Men W, Pre < 4, Day 6: number analyzed (Participants) | 31 | 28 | 59 | 16
  hSBA-Men W, Pre < 4, Day 6 | 64.52 [45.37 to 80.77] | 75 [55.13 to 89.31] | 69.49 [56.13 to 80.81] | 25 [7.27 to 52.38]
  hSBA-Men W, Pre ≥ 4, Day 6: number analyzed (Participants) | 114 | 112 | 226 | 28
  hSBA-Men W, Pre ≥ 4, Day 6 | 46.49 [37.1 to 56.07] | 42.86 [33.55 to 52.55] | 44.69 [38.09 to 51.43] | 3.57 [0.09 to 18.35]
  hSBA-Men W, Total seroresponse, Day 6: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men W, Total seroresponse, Day 6 | 50.34 [41.93 to 58.75] | 49.29 [40.74 to 57.86] | 49.82 [43.87 to 55.78] | 11.36 [3.79 to 24.56]
  hSBA-Men Y, Pre < 4, Day 4: number analyzed (Participants) | 62 | 60 | 122 | 27
  hSBA-Men Y, Pre < 4, Day 4 | 8.06 [2.67 to 17.83] | 6.67 [1.85 to 16.2] | 7.38 [3.43 to 13.54] | 0 [0 to 12.77]
  hSBA-Men Y, Pre ≥ 4, Day 4: number analyzed (Participants) | 80 | 77 | 157 | 21
  hSBA-Men Y, Pre ≥ 4, Day 4 | 7.5 [2.8 to 15.61] | 2.6 [0.32 to 9.07] | 5.1 [2.23 to 9.79] | 0 [0 to 16.11]
  hSBA-Men Y, Total seroresponse, Day 4: number analyzed (Participants) | 142 | 137 | 279 | 48
  hSBA-Men Y, Total seroresponse, Day 4 | 7.75 [3.93 to 13.44] | 4.38 [1.62 to 9.29] | 6.09 [3.59 to 9.58] | 0 [0 to 7.4]
  hSBA-Men Y, Pre < 4, Day 6: number analyzed (Participants) | 52 | 62 | 114 | 27
  hSBA-Men Y, Pre < 4, Day 6 | 63.46 [48.96 to 76.38] | 75.81 [63.26 to 85.78] | 70.18 [60.89 to 78.38] | 11.11 [2.35 to 29.16]
  hSBA-Men Y, Pre ≥ 4, Day 6: number analyzed (Participants) | 91 | 78 | 169 | 17
  hSBA-Men Y, Pre ≥ 4, Day 6 | 40.66 [30.48 to 51.47] | 42.31 [31.19 to 54.02] | 41.42 [33.91 to 49.24] | 5.88 [0.15 to 28.69]
  hSBA-Men Y, Total seroresponse, Day 6: number analyzed (Participants) | 143 | 140 | 283 | 44
  hSBA-Men Y, Total seroresponse, Day 6 | 48.95 [40.51 to 57.44] | 57.14 [48.51 to 65.47] | 53 [47.01 to 58.94] | 9.09 [2.53 to 21.67]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- Day 4- Total seroresponse (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 1.39, 95% CI 2-sided [-6.08 to 4.94]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- Day 4-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 2.17, 95% CI 2-sided [-5.32 to 6.21]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- Day 4-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 1.77, 95% CI 2-sided [-5.68 to 4.09]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- Day 4-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -0.79, 95% CI 2-sided [-4.98 to 3.01]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A- Day 6-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 34.76, 95% CI 2-sided [22.38 to 44.07]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A- Day 6-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 26.88, 95% CI 2-sided [14.67 to 36.13]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A- Day 6-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 30.89, 95% CI 2-sided [19.42 to 37.97]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A- Day 6-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 7.88, 95% CI 2-sided [-3.25 to 18.81]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- Day 4-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -3.45, 95% CI 2-sided [-14.26 to 2.35]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- Day 4-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 2.51, 95% CI 2-sided [-8.70 to 9.98]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- Day 4-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -0.54, 95% CI 2-sided [-11.35 to 4.90]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- Day 4-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -5.96, 95% CI 2-sided [-12.25 to -0.57]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C- Day 6-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 40.03, 95% CI 2-sided [25.37 to 50.92]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C- Day 6-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 36.84, 95% CI 2-sided [22.14 to 47.90]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C- Day 6-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 38.46, 95% CI 2-sided [24.79 to 47.57]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C- Day 6-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 3.19, 95% CI 2-sided [-8.44 to 14.73]
Statistical Analysis 17: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- Day 4-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -3.47, 95% CI 2-sided [-14.28 to 2.31]
Statistical Analysis 18: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- Day 4-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 3.89, 95% CI 2-sided [-7.40 to 11.60]
Statistical Analysis 19: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- Day 4-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 0.13, 95% CI 2-sided [-10.70 to 5.66]
Statistical Analysis 20: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- Day 4-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -7.37, 95% CI 2-sided [-13.89 to -1.80]
Statistical Analysis 21: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W- Day 6-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 38.98, 95% CI 2-sided [24.35 to 49.88]
Statistical Analysis 22: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W- Day 6-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 37.92, 95% CI 2-sided [23.23 to 48.95]
Statistical Analysis 23: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W- Day 6-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 38.46, 95% CI 2-sided [24.80 to 47.56]
Statistical Analysis 24: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W- Day 6-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 1.06, 95% CI 2-sided [-10.51 to 12.60]
Statistical Analysis 25: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- Day 4-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 7.75, 95% CI 2-sided [0.15 to 13.36]
Statistical Analysis 26: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- Day 4-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 4.38, 95% CI 2-sided [-3.15 to 9.24]
Statistical Analysis 27: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- Day 4-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 6.09, 95% CI 2-sided [-1.41 to 9.55]
Statistical Analysis 28: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- Day 4-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 3.37, 95% CI 2-sided [-2.48 to 9.54]
Statistical Analysis 29: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y- Day 6-Total seroresponse- (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 39.86, 95% CI 2-sided [25.76 to 50.29]
Statistical Analysis 30: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y- Day 6-Total seroresponse - (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 48.05, 95% CI 2-sided [33.89 to 58.34]
Statistical Analysis 31: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y- Day 6-Total seroresponse - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = 43.91, 95% CI 2-sided [30.79 to 52.37]
Statistical Analysis 32: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y- Day 6-Total seroresponse - (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 1, analysis 1]; Miettinen & Nurminen score method; Differences in percentage = -8.19, 95% CI 2-sided [-19.61 to 3.45]

16. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroup A, C, W and Y.
Description: For each N. meningitidis serogroup A, C, W and Y, unadjusted GMTs were calculated, with their associated two-sided 95% Confidence Interval.
Time Frame: At Day 1 (pre-vaccination), Day 4, Day 6 and Day 29
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 290 | 282 | 572 | 93
Titers
  hSBA-Men A, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men A, Day 1 | 2.81 [2.54 to 3.11] | 2.95 [2.67 to 3.27] | 2.88 [2.68 to 3.09] | 2.27 [1.9 to 2.71]
  hSBA-Men A, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men A, Day 4 | 2.83 [2.43 to 3.29] | 3 [2.57 to 3.51] | 2.91 [2.61 to 3.25] | 2.25 [1.73 to 2.93]
  hSBA-Men A, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men A, Day 6 | 12.87 [9.63 to 17.19] | 10.17 [7.57 to 13.66] | 11.47 [9.32 to 14.1] | 2.48 [1.46 to 4.2]
  hSBA-Men A, Day 29 | 210.1 [181.07 to 243.78] | 236.69 [203.56 to 275.2] | 222.81 [200.43 to 247.7] | 32.11 [24.7 to 41.76]
  hSBA-Men C, Day 1: number analyzed (Participants) | 288 | 281 | 569 | 93
  hSBA-Men C, Day 1 | 16.11 [13.28 to 19.54] | 10.72 [8.82 to 13.03] | 13.17 [11.48 to 15.12] | 5.06 [3.6 to 7.1]
  hSBA-Men C, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men C, Day 4 | 22.96 [17.31 to 30.45] | 14.29 [10.71 to 19.07] | 18.21 [14.86 to 22.31] | 6.69 [4.1 to 10.9]
  hSBA-Men C, Day 6: number analyzed (Participants) | 145 | 139 | 284 | 44
  hSBA-Men C, Day 6 | 92.27 [68.91 to 123.56] | 90.06 [66.84 to 121.35] | 91.18 [74.04 to 112.3] | 6.71 [3.95 to 11.4]
  hSBA-Men C, Day 29: number analyzed (Participants) | 290 | 281 | 571 | 93
  hSBA-Men C, Day 29 | 1159.93 [977.33 to 1376.63] | 1057.66 [888.74 to 1258.68] | 1108.42 [981.09 to 1252.27] | 59.7 [44.12 to 80.78]
  hSBA-Men W, Day 1: number analyzed (Participants) | 289 | 282 | 571 | 93
  hSBA-Men W, Day 1 | 22.07 [18.54 to 26.29] | 23.46 [19.66 to 28] | 22.75 [20.09 to 25.76] | 12.21 [8.98 to 16.62]
  hSBA-Men W, Day 4: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men W, Day 4 | 25.9 [20.13 to 33.32] | 33.87 [26.18 to 43.82] | 29.53 [24.66 to 35.37] | 13.8 [8.92 to 21.35]
  hSBA-Men W, Day 6: number analyzed (Participants) | 146 | 140 | 286 | 44
  hSBA-Men W, Day 6 | 112.49 [86.26 to 146.71] | 143.75 [109.61 to 188.54] | 126.84 [104.9 to 153.37] | 15.98 [9.85 to 25.93]
  hSBA-Men W, Day 29: number analyzed (Participants) | 290 | 281 | 571 | 92
  hSBA-Men W, Day 29 | 1394.65 [1176.59 to 1653.11] | 1883.96 [1585.12 to 2239.15] | 1617.11 [1431.93 to 1826.23] | 55.31 [40.9 to 74.8]
  hSBA-Men Y, Day 1: number analyzed (Participants) | 287 | 281 | 568 | 93
  hSBA-Men Y, Day 1 | 9.24 [7.81 to 10.94] | 8.22 [6.93 to 9.75] | 8.72 [7.74 to 9.83] | 4.56 [3.39 to 6.13]
  hSBA-Men Y, Day 4: number analyzed (Participants) | 143 | 138 | 281 | 48
  hSBA-Men Y, Day 4 | 10.87 [8.26 to 14.32] | 12.12 [9.16 to 16.04] | 11.47 [9.43 to 13.95] | 4.63 [2.88 to 7.44]
  hSBA-Men Y, Day 6: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men Y, Day 6 | 63.3 [47.73 to 83.95] | 61.56 [46.18 to 82.05] | 62.44 [51.06 to 76.34] | 6.44 [3.86 to 10.76]
  hSBA-Men Y, Day 29: number analyzed (Participants) | 290 | 281 | 571 | 93
  hSBA-Men Y, Day 29 | 1066.66 [900.67 to 1263.25] | 1007.62 [848.53 to 1196.54] | 1037.19 [919.46 to 1169.98] | 37.4 [27.75 to 50.42]
Statistical Analysis 1: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 4(Menveo-Menveo vs. Naive); Test type: Other — GMTs ratio and 95% CI, at each time point against each serogroups A, C, W and Y strains was obtained by exponentiating the mean between-group differences in log-transformed titers and the corresponding 95% CIs at each of the timepoints specified; Between group GMT ratios = 1.26, 95% CI 2-sided [0.93 to 1.70]
Statistical Analysis 2: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 4(Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.34, 95% CI 2-sided [0.98 to 1.82]
Statistical Analysis 3: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A-Vaccine comparison at day 4(Pooled Menveo-Menveo and Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.29, 95% CI 2-sided [0.97 to 1.72]
Statistical Analysis 4: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A-Vaccine comparison at day 4 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.94, 95% CI 2-sided [0.76 to 1.17]
Statistical Analysis 5: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 6 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 5.19, 95% CI 2-sided [2.84 to 9.47]
Statistical Analysis 6: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 6 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 4.10, 95% CI 2-sided [2.24 to 7.50]
Statistical Analysis 7: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A-Vaccine comparison at day 6 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 4.62, 95% CI 2-sided [2.62 to 8.15]
Statistical Analysis 8: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A-Vaccine comparison at day 6 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.27, 95% CI 2-sided [0.84 to 1.91]
Statistical Analysis 9: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 29 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 6.54, 95% CI 2-sided [4.84 to 8.85]
Statistical Analysis 10: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup A-Vaccine comparison at day 29 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 7.37, 95% CI 2-sided [5.44 to 9.98]
Statistical Analysis 11: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup A-Vaccine comparison at day 29 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 6.94, 95% CI 2-sided [5.23 to 9.21]
Statistical Analysis 12: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup A-Vaccine comparison at day 29 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.89, 95% CI 2-sided [0.72 to 1.10]
Statistical Analysis 13: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 4 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; between group GMT ratios = 3.43, 95% CI 2-sided [1.95 to 6.04]
Statistical Analysis 14: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 4 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.14, 95% CI 2-sided [1.21 to 3.77]
Statistical Analysis 15: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C-Vaccine comparison at day 4 - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.72, 95% CI 2-sided [1.60 to 4.64]
Statistical Analysis 16: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C-Vaccine comparison at day 4 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.61, 95% CI 2-sided [1.07 to 2.40]
Statistical Analysis 17: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 6 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 13.75, 95% CI 2-sided [7.51 to 25.19]
Statistical Analysis 18: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 6 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 13.42, 95% CI 2-sided [7.31 to 24.66]
Statistical Analysis 19: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C-Vaccine comparison at day 6 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 13.59, 95% CI 2-sided [7.70 to 24.00]
Statistical Analysis 20: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C-Vaccine comparison at day 6 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.02, 95% CI 2-sided [0.67 to 1.56]
Statistical Analysis 21: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 29 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 19.43, 95% CI 2-sided [13.73 to 27.51]
Statistical Analysis 22: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup C-Vaccine comparison at day 29 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 17.72, 95% CI 2-sided [12.50 to 25.12]
Statistical Analysis 23: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup C-Vaccine comparison at day 29 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 18.57, 95% CI 2-sided [13.40 to 25.73]
Statistical Analysis 24: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup C-Vaccine comparison at day 29 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.10, 95% CI 2-sided [0.86 to 1.40]
Statistical Analysis 25: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 4 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.88, 95% CI 2-sided [1.13 to 3.11]
Statistical Analysis 26: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 4 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.46, 95% CI 2-sided [1.48 to 4.08]
Statistical Analysis 27: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W-Vaccine comparison at day 4 - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.14, 95% CI 2-sided [1.33 to 3.44]
Statistical Analysis 28: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W-Vaccine comparison at day 4 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.76, 95% CI 2-sided [0.53 to 1.10]
Statistical Analysis 29: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 6 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 7.04, 95% CI 2-sided [4.05 to 12.22]
Statistical Analysis 30: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 6 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 8.99, 95% CI 2-sided [5.16 to 15.66]
Statistical Analysis 31: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W-Vaccine comparison at day 6 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 7.94, 95% CI 2-sided [4.72 to 13.35]
Statistical Analysis 32: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W-Vaccine comparison at day 6 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.78, 95% CI 2-sided [0.54 to 1.14]
Statistical Analysis 33: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 29 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 25.21, 95% CI 2-sided [17.83 to 35.65]
Statistical Analysis 34: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup W-Vaccine comparison at day 29 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 34.06, 95% CI 2-sided [24.06 to 48.23]
Statistical Analysis 35: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup W-Vaccine comparison at day 29 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 29.24, 95% CI 2-sided [21.09 to 40.52]
Statistical Analysis 36: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup W-Vaccine comparison at day 29 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.74, 95% CI 2-sided [0.58 to 0.94]
Statistical Analysis 37: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 4 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.35, 95% CI 2-sided [1.36 to 4.07]
Statistical Analysis 38: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 4 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.62, 95% CI 2-sided [1.51 to 4.54]
Statistical Analysis 39: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y-Vaccine comparison at day 4 - (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 2.48, 95% CI 2-sided [1.48 to 4.14]
Statistical Analysis 40: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y-Vaccine comparison at day 4 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 0.90, 95% CI 2-sided [0.61 to 1.33]
Statistical Analysis 41: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 6 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 9.82, 95% CI 2-sided [5.47 to 17.64]
Statistical Analysis 42: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 6 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 9.55, 95% CI 2-sided [5.31 to 17.19]
Statistical Analysis 43: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y-Vaccine comparison at day 6 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 9.69, 95% CI 2-sided [5.59 to 16.79]
Statistical Analysis 44: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y-Vaccine comparison at day 6 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.03, 95% CI 2-sided [0.69 to 1.54]
Statistical Analysis 45: Comparison: Menveo-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 29 (Menveo-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 28.52, 95% CI 2-sided [20.23 to 40.20]
Statistical Analysis 46: Comparison: Menactra-Menveo Group vs Naive Group; Serogroup Y-Vaccine comparison at day 29 (Menactra-Menveo vs. Naive); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 26.94, 95% CI 2-sided [19.09 to 38.02]
Statistical Analysis 47: Comparison: Pooled Group (Menveo-Menveo and Menactra-Menveo) vs Naive Group; Serogroup Y-Vaccine comparison at day 29 (Pooled Menveo-Menveo and Menactra-Menveo vs. Naïve); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 27.73, 95% CI 2-sided [20.10 to 38.26]
Statistical Analysis 48: Comparison: Menveo-Menveo Group vs Menactra-Menveo Group; Serogroup Y-Vaccine comparison at day 29 (Menveo-Menveo vs. Menactra-Menveo); Test type: Other — [test comment as in outcome 16, analysis 1]; Between group GMT ratios = 1.06, 95% CI 2-sided [0.83 to 1.35]

17. Secondary Outcome: Within Group hSBA Geometric Mean Ratios (GMRs)
Description: Within each study group and for each serogroup, GMRs were calculated,at: Visit Day 4 versus at Visit Day 1; Visit Day 6 versus at Visit Day 1; and Visit Day 29 versus at Visit Day 1. The unadjusted GMRs and 95% CIs are constructed by exponentiating the mean within-group differences in log-transformed titers and the corresponding 95% CIs.
Time Frame: At Day 4, Day 6, Day 29 compared to Day 1
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Pooled Group (Menveo-Menveo and Menactra-Menveo) | Naive Group
Number analyzed (Participants) | 289 | 282 | 571 | 93
Ratios
  hSBA-Men A, Day 4/Day 1: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men A, Day 4/Day 1 | 1.02 [0.93 to 1.12] | 1.07 [0.97 to 1.17] | 1.04 [0.98 to 1.11] | 0.99 [0.84 to 1.16]
  hSBA-Men A, Day 6/Day 1: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men A, Day 6/Day 1 | 4.58 [3.49 to 6] | 3.25 [2.46 to 4.28] | 3.87 [3.19 to 4.7] | 1.09 [0.66 to 1.78]
  hSBA-Men A, Day 29/Day 1 | 75.02 [63.87 to 88.12] | 80.13 [68.09 to 94.3] | 77.5 [69.12 to 86.9] | 14.14 [10.65 to 18.77]
  hSBA-Men C, Day 4/Day 1: number analyzed (Participants) | 143 | 137 | 280 | 48
  hSBA-Men C, Day 4/Day 1 | 1.12 [0.99 to 1.28] | 1.35 [1.19 to 1.54] | 1.23 [1.12 to 1.35] | 1.21 [0.97 to 1.51]
  hSBA-Men C, Day 6/Day 1: number analyzed (Participants) | 144 | 139 | 283 | 44
  hSBA-Men C, Day 6/Day 1 | 7.25 [5.39 to 9.75] | 7.94 [5.87 to 10.73] | 7.58 [6.14 to 9.36] | 1.45 [0.85 to 2.48]
  hSBA-Men C, Day 29/Day 1: number analyzed (Participants) | 288 | 280 | 568 | 93
  hSBA-Men C, Day 29/Day 1 | 71.72 [58.88 to 87.37] | 97.13 [79.51 to 118.65] | 83.29 [72.34 to 95.89] | 11.81 [8.34 to 16.71]
  hSBA-Men W, Day 4/Day 1: number analyzed (Participants) | 144 | 138 | 282 | 48
  hSBA-Men W, Day 4/Day 1 | 1.05 [0.91 to 1.23] | 1.4 [1.2 to 1.63] | 1.21 [1.09 to 1.35] | 1.14 [0.88 to 1.48]
  hSBA-Men W, Day 6/Day 1: number analyzed (Participants) | 145 | 140 | 285 | 44
  hSBA-Men W, Day 6/Day 1 | 5.71 [4.37 to 7.45] | 6.27 [4.78 to 8.23] | 5.98 [4.95 to 7.23] | 1.32 [0.81 to 2.15]
  hSBA-Men W, Day 29/Day 1: number analyzed (Participants) | 289 | 281 | 570 | 92
  hSBA-Men W, Day 29/Day 1 | 63.63 [51.37 to 78.81] | 80.61 [64.88 to 100.14] | 71.5 [61.38 to 83.27] | 4.57 [3.13 to 6.68]
  hSBA-Men Y, Day 4/Day 1: number analyzed (Participants) | 142 | 137 | 279 | 48
  hSBA-Men Y, Day 4/Day 1 | 1.35 [1.15 to 1.59] | 1.31 [1.11 to 1.54] | 1.33 [1.19 to 1.49] | 0.99 [0.75 to 1.31]
  hSBA-Men Y, Day 6/Day 1: number analyzed (Participants) | 143 | 140 | 283 | 44
  hSBA-Men Y, Day 6/Day 1 | 6.09 [4.53 to 8.19] | 8.59 [6.37 to 11.59] | 7.22 [5.85 to 8.92] | 1.48 [0.87 to 2.52]
  hSBA-Men Y, Day 29/Day 1: number analyzed (Participants) | 287 | 280 | 567 | 93
  hSBA-Men Y, Day 29/Day 1 | 116.58 [94.42 to 143.95] | 123.41 [99.69 to 152.78] | 119.91 [103.21 to 139.3] | 8.21 [5.67 to 11.89]

ADVERSE EVENTS:
Time Frame: Solicited AEs were assessed between 6 hours through Day 7. Unsolicited AEs were assessed between Day 1 trough Day 29. SAEs were assessed during the entire study period (from Day 1 to Day 181).
Arm/Group | Menveo-Menveo Group | Menactra-Menveo Group | Naive Group
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/300 | 0/100
Serious Adverse Events (participants affected / at risk) | 3/301 | 2/300 | 3/100
Other Adverse Events (participants affected / at risk) | 243/301 | 211/300 | 60/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menveo-Menveo Group (N=301) | Menactra-Menveo Group (N=300) | Naive Group (N=100)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menveo-Menveo Group (N=301) | Menactra-Menveo Group (N=300) | Naive Group (N=100)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Oculogyric crisis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 51 (65) | 44 (55) | 15 (17)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland mucocoele (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 119 (124) | 106 (113) | 41 (41)
Fatigue (General disorders) | 116 (146) | 111 (159) | 19 (21)
Chills (General disorders) | 34 (36) | 37 (50) | 10 (10)
Injection site induration (General disorders) | 17 (17) | 10 (11) | 8 (9)
Injection site erythema (General disorders) | 14 (16) | 10 (10) | 11 (14)
Pyrexia (General disorders) | 3 (4) | 7 (8) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 2 (2) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (16) | 5 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 9 (9) | 3 (3)
Acute sinusitis (Infections and infestations) | 11 (13) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 7 (7) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Viral pharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 6 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (4)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 6 (6) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 37 (50) | 48 (63) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 57 (63) | 55 (72) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 (60) | 41 (50) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 103 (135) | 84 (118) | 23 (27)
Syncope (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphangiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT02986854/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT02986854/SAP_001.pdf